CLINICAL TRIAL: NCT04712708
Title: Role of Rebound Therapy in the Rehabilitation of Children With Spastic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Faten Hassan Abdelaziem, Prof . Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T. REC/012/002421
Record Dates: First submitted 2021-01-04; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Eighteen children with spastic CP will receive especially designed physical therapy program based on Neuro-Developmental treatment (NDT) approach with emphasis on exercise encourage independent standing, stretches exercises, strengthening exercises, approximation, enhancement and facilitation of gait patterning and ankle ROM exercises for one hour for 24 sessions
  Interventions: Other: Physical Therapy Program
- Study Group (Experimental): ighteen children with spastic CP will receive the same program that the control group received in addition to especially designed exercises using rebound therapy (Mini Trampoline) that include push up exercise, standing, squatting, single limb squatting, kneeling position, catching and throwing a ball over head in kneeling position, catching and throwing a ball over head in standing position, kicking the ball, broad jumping with assistance, jumping in place, for 1 hour three times per week for three successive months.
  Interventions: Device: Rebound Therapy; Other: Physical Therapy Program

INTERVENTIONS:
Device: Rebound Therapy — Rebound therapy is the therapeutic use of full sized trampoline or mini sized trampoline. It provides opportunities for exercise recreation and therapy; and it is distinct from gymnastic trampolining. It is used for facilitating movements, improving balance, enhancing coordination and promoting motor performances in children with different disorders includes learning disabilities, communication disorders and motor dysfunction (Rebound Therapy South Africa, 2020; The Chartered society of Physiotherapists, 2016).
  Arms: Study Group
Other: Physical Therapy Program — The Mat Exercises:
  Stretching exercises to all spastic muscle groups (Kalkman et al., 2018). Gentle exercises was applied for 40-60 seconds and repeated from 3-5 times/ movement as supported by (Fragala et al., 2003).
  Strengthening Exercises:
  Dynamic Rising Positioning
  The Gym Exercises:

SUMMARY:
Cerebral palsy (CP) is a group of disorders of movement and posture, causing several body impairments. CP is caused by non-progressive disturbance that occurred in the fetal or immature brain. CP symptoms include several motor disorders such as disturbances in sensation, coordination, cognition, communication and behavior in addition to disturbances in postural stability, balance and coordination.

Balance is the ability to maintain the center of body mass over the base of support. CP causes balance impairment which results in decrease in the child's mobility functions and causing activity limitation and participations restrictions.

Motor coordination is the registration of two or more things such as body movements , timing or sensory feedback into a harmonious relationship.

CP causes disturbances in motor coordination such as difficulties in the routine gross movements as running and jumping, and disturbances in common fine movements like buttoning, clothing or brushing hair Rebound therapy is an exercise therapy which uses mini trampolines, rebounders , Springfree Trampoline and Swiss balls, to provide opportunity to perform recreational movements for individuals with different body structural and functional impairments.

ELIGIBILITY:
Inclusion Criteria:

* Spastic cerebral palsy was determined according to the sample size calculation, was selected from the outpatient's clinic of the faculty of Physical Therapy Cairo University.
* Level I according to the Gross Motor Function Classification System (GMFCS). Chronological age ranged from 5 to 11 years.
* Height was above 1 meter.
* Understand verbal command.
* The degree of spasticity ranged from 1 to 1+ according to Modified Ashworth' Scale.

Rebound therapy using trampoline was used as the method of management in the study group in addition to the selected physical therapy program that was used in both groups, and the treatment sessions was provided in the out-patient clinic of the faculty of Physical Therapy Cairo University.

Exclusion Criteria:

* Vertigo or dizziness.
* Epilepsy.
* Osteoporosis.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Balance | 12 Weeks
  Stationary Balance Using Biodex Balance System
Gross Motor Function | 12 Weeks
  Gross Motor Function using Gross Motor Function Measure (GMFM)
Gross Motor Coordination | 12 Weeks
  Gross Motor Coordination Using Gross Motor Coordination Quotient in BOT-2

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided